CLINICAL TRIAL: NCT07293975
Title: Assessment of Transcutaneous Electrical Nerve Stimulation and High-Frequency Vibration for Pain Control During Bracket Debonding: A Clinical Trial Study
Brief Title: Pain Control During Braces Removal Using Transcutaneous Electrical Nerve Stimulation and High-Frequency Vibration
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Malak Ramzi Abdulmoula Alsaqqaf, Student Researcher, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TENS-VIB-PAIN-2025
Record Dates: First submitted 2025-12-09; First posted 2025-12-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Orthodontic Pain
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups: TENS, high-frequency vibration, or control. Each participant will undergo a single session in which the assigned intervention is applied. The study is open-label, and all bracket removal procedures are performed by the same operator using standardized techniques to ensure consistency across groups. Baseline dental anxiety and sex will be recorded as covariates for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Transcutaneous Electrical Nerve Stimulation (TENS) (Experimental): Participants in this arm will receive transcutaneous electrical nerve stimulation (TENS) applied immediately before orthodontic bracket removal. Pain, satisfaction, and procedural efficiency will be assessed during a single session.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- High-Frequency Vibration (SureSmile® VPro™) (Experimental): Participants in this arm will receive high-frequency vibration applied during orthodontic bracket removal. Pain, satisfaction, and procedural efficiency will be assessed during a single session.
  Interventions: Device: High-Frequency Vibration
- No Intervention (No Intervention): Participants in this arm will undergo standard orthodontic bracket removal without any additional device. Pain, satisfaction, and procedural efficiency will be assessed during a single session.

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — TENS is applied immediately before orthodontic bracket removal in a single session to reduce pain and improve patient satisfaction.
  Arms: Transcutaneous Electrical Nerve Stimulation (TENS)
Device: High-Frequency Vibration — High-frequency vibration is applied during orthodontic bracket removal in a single session to reduce pain and improve patient satisfaction.
  Arms: High-Frequency Vibration (SureSmile® VPro™)

SUMMARY:
This study aims to find the best method to reduce pain during braces removal. We are comparing transcutaneous electrical nerve stimulation (TENS), high-frequency vibration, and a control group with no additional intervention.

People who have completed orthodontic treatment and need their braces removed can take part. Participants will be randomly assigned to one of the three groups. The vibration device will be applied during the braces removal, while TENS will be applied just before the procedure.

Before the procedure, participants' anxiety will be measured using the Modified Dental Anxiety Scale (MDAS). During and after the procedure, pain will be assessed using a Visual Analog Scale (VAS) from 0 to 100, and participants will rate their satisfaction using a Numerical Rating Scale (NRS) from 0 to 10.

The purpose of this research is to help orthodontists identify the method that makes braces removal less uncomfortable, more tolerable, and more satisfying for patients.

DETAILED DESCRIPTION:
This clinical study aims to evaluate and compare the effectiveness and cost-effectiveness of TENS (Dental Pain Eraser) and high-frequency vibration (SureSmile® VPro™) in reducing discomfort during orthodontic bracket removal, improving patient satisfaction, and optimizing efficiency. The study includes a control group, and results are intended to provide evidence-based guidance for orthodontists to enhance the patient experience during debonding procedures.

Participants will be individuals who have completed fixed orthodontic treatment and are scheduled for bracket removal. Before the procedure, their baseline dental anxiety will be assessed. The assigned intervention will be applied either immediately before (TENS) or during (vibration) the bracket removal session. Participants' experiences of pain and satisfaction will be monitored throughout the procedure. Sex and baseline anxiety will be considered in the analysis to evaluate their influence on outcomes. A cost-effectiveness analysis will be performed to determine the most efficient method among the interventions.

The research will be conducted in a standardized clinical setting, adhering to established bracket removal protocols to ensure participant safety and minimize variability. The procedures will be performed by the same operator following consistent techniques.

This study is designed to generate practical insights into pain management during orthodontic debonding, focusing on participant comfort, satisfaction, and procedural efficiency, without compromising the quality of care. The findings may guide future clinical recommendations and improve patient-centered orthodontic practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for fixed orthodontic appliance removal.
2. Permanent dentition present, including both anterior and posterior teeth.
3. Age between 15-35 years.
4. Ability to provide informed consent and comply with study procedures.
5. General health adequate for routine orthodontic care.
6. No history of regular or recent medication intake within the preceding 24 hours, including painkillers, corticosteroids, or anti-flu drugs.

Exclusion Criteria:

1. Patients with craniofacial anomalies, systemic conditions affecting pain perception, or taking medications influencing nociception.
2. Teeth with extensive restorations or prostheses that prevent standard bracket debonding.
3. Patients with known allergy or contraindication to TENS or vibration devices.
4. Pregnant women.
5. Active periodontal disease, including gingival recession or tooth mobility exceeding Grade I.
6. Excessive gingival overgrowth that may impede debonding or influence study outcomes.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pain During Orthodontic Debonding Measured by VAS | During and immediately after debonding procedure
  Pain during debonding will be measured immediately after the procedure using VAS 0-100 mm, where 0 = no pain and 100 = worst imaginable pain.

SECONDARY OUTCOMES:
Baseline Anxiety | Prior to the debonding procedure
  Baseline anxiety will be assessed prior to the debonding procedure using the Modified Dental Anxiety Scale (MDAS).
  The MDAS consists of five items, each scored on a 5-point Likert scale as follows:
  Not anxious = 1; Slightly anxious = 2; Fairly anxious = 3; Very anxious = 4; Extremely anxious = 5.
  The total MDAS score is calculated as the sum of all five items, with a possible range from 5 to 25.
  A cut-off score of 19 or above indicates a highly dentally anxious patient, possibly dentally phobic.
  Higher scores indicate greater dental anxiety (worse outcome).
Patient Satisfaction | immediately post-procedure
  Satisfaction will be assessed immediately post-procedure using Numeric Rating Scale (0-10) to evaluate comfort and overall acceptance of the method.
Device Application Time | Periprocedural (during the debonding session)
  Device application time will be recorded for each intervention and defined as the duration (in seconds) required to apply the pain reduction method prior to and/or during orthodontic debonding.
Cost-Effectiveness Analysis | Periprocedural (during the debonding session) and at immediate post-procedure assessment.
  Direct costs, including device cost, consumables, and operator time, will be recorded for each intervention.
  Cost-effectiveness ratios will be calculated as cost per unit reduction in pain score (VAS) to compare the efficiency of each pain-reduction method.

CONTACTS AND LOCATIONS:
Overall Officials: Ali M. Al-Attar, BDS, MSc, PhD, Principal Investigator — University of Baghdad - College of Dentistry - Orthodontics

IPD SHARING:
Plan to Share IPD: No
There is currently no definitive plan to share Individual Participant Data (IPD). However, IPD may be made available in the future if required by the journal in which the results are published, subject to ethical approval, institutional regulations, and obtaining appropriate patient consent. All shared data will be de-identified to protect participant confidentiality.